Clinical Trials 9/26/19
Internet-based videoconferencing to address alcohol use and pain among heavy drinkers in HIV-care
NCT03982433

## Summary:

Open pilot trial of 8 patients in HIV care. All patients screened were assigned to the intervention condition with the goal of assessing acceptability and feasibility.

Descriptive analyses only for this acceptability and feasibility study Mean and median ratings as pre-specified for primary outcomes

## **Procedures**

Participants were screened by phone or in-person. Eligible participants were scheduled to complete the initial visit that consisted of consent procedures, a 50-minute baseline assessment, followed by an initial in-person session with a clinical psychologist. The initial in-person session provided a rationale for the program and established technology procedures for the subsequent video-conferencing intervention (e.g., downloading the app, receiving the session link, etc.). Prior to leaving the initial session, participants practiced videoconferencing using their own smartphones. Participants were scheduled to complete the first videoconferencing session within a week of the baseline interview. Subsequent sessions were scheduled weekly for a total of 6 video-conferencing sessions.

To facilitate engagement, participants were reminded via text message the day before and the day of the intervention. Five minutes prior to the appointment time, they were sent a link for the videoconferencing meeting either by text or via email. Those who experienced any difficulties using the technology were able to consult the "troubleshooting" form that they were given or call the study assistant who could guide them through the videoconferencing procedures. Videoconferencing sessions were scheduled for up to 45 minutes and ranged from 20-45 minutes depending on the topic and the participant. Each videoconferencing session began with a review of symptoms and review of skills used in the previous week followed by the topic for the current

week. In addition to the live session with the interventionist, participants were also sent brief (2-minute) video demonstrations for some of the skills that they learned and worksheets to remind them of content and homework through a secure app. Participants were permitted to reschedule up to 3 sessions; more than 3 sessions counted as missed appointments. The post-intervention assessment was conducted in person by a research assistant approximately 8 weeks after the baseline interview.

## Analysis Plan

Descriptive analyses of self-report and behavioral outcomes were performed using SPSS v. 24. Number of videoconferencing sessions attended (out of 6) for all participants were recorded. Post-intervention assessments were available from 7 of the 8 participants in the study. Means, standard deviations and medians were calculated for continuous variables and count data. Median pain severity and interference as well as number of heavy drinking days and drinks per week were examined as the primary symptom variables in addition to self-report measures of self-regulatory skills related to pain management and alcohol use.